CLINICAL TRIAL: NCT02205047
Title: INtegratioN of Trastuzumab, With or Without Pertuzumab, Into periOperatiVe chemotherApy of HER-2 posiTIve stOmach caNcer: the INNOVATION-TRIAL
Brief Title: Neoadjuvant Study Using Trastuzumab or Trastuzumab With Pertuzumab in Gastric or Gastroesophageal Junction Adenocarcinoma
Acronym: INNOVATION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1203-GITCG; 2014-000722-38 (EudraCT Number); MO28922 (Other Grant/Funding Number: Roche)
Record Dates: First submitted 2014-07-10; First posted 2014-07-31 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Malignant Neoplasm of Stomach; Malignant Neoplasm of Cardio-esophageal Junction of Stomach; Epidermal Growth Factor Receptor (EGFR) Protein Overexpression
Keywords: Neoadjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Fluorouracil; Capecitabine; Trastuzumab; pertuzumab; Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard chemotherapy (Active Comparator): Cisplatin/capecitabine or cisplatin/5-fluorouracil
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil or Capecitabine; Procedure: gastrectomy
- Experimental arm 1 (Experimental): Cisplatin/capecitabine plus trastuzumab or cisplatin/5-fluorouracil plus trastuzumab
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil or Capecitabine; Drug: Trastuzumab; Procedure: gastrectomy
- Experimental arm 2 (Experimental): cisplatin/capecitabine plus trastuzumab and pertuzumab or cisplatin/5-fluorouracil plus trastuzumab and pertuzumab
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil or Capecitabine; Drug: Trastuzumab; Drug: Pertuzumab; Procedure: gastrectomy

INTERVENTIONS:
Drug: Cisplatin
Drug: 5-fluorouracil or Capecitabine
Drug: Trastuzumab
  Arms: Experimental arm 1; Experimental arm 2
Drug: Pertuzumab
  Arms: Experimental arm 2
Procedure: gastrectomy — D2 gastrectomy

SUMMARY:
The purpose of this study is to find out whether either trastuzumab or the combination of trastuzumab and pertuzumab with standard chemotherapy shows more activity against gastro-oesophageal adenocarcinoma than standard chemotherapy given before and after surgery and it can be safely administered.

DETAILED DESCRIPTION:
This is a randomized phase II trial with an internal control. The randomization will be a 1:2:2 randomization (control: experimental arm 1: experimental arm 2). Potentially eligible patients will be screened centrally for the HER-2 status. After confirmation of HER-2 positive disease, eligible patients will be centrally randomized through the EORTC randomization system. A minimization technique will be used for random treatment allocation between the three treatment arms. Stratification will be done by histological subtype (intestinal/non-intestinal); Korea versus Europe; stage II versus III; node positive versus node negative.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, gastric or gastroesophageal (GE)-junction adenocarcinoma (Siewert I-III)
* Patient medically fit for gastrectomy/oesophagogastrectomy as decided by the investigator
* Age ≥ 18 years
* WHO performance status 0 - 1
* HER-2 overexpression
* Amenable to gastrectomy/oesophagectomy
* The cardiac ejection fraction (LVEF), as determined by echocardiography, multiple gated acquisition scan (MUGA) or cardiac MRI should be at least 50 %
* Adequate organ function
* written informed consent
* For women who are not postmenopausal (> 12 months of non-therapy induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 12 months after the last treatment dose
* For men: agreement to remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 12 months after the last dose of study treatment. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods for contraception.

Exclusion Criteria:

* Absence of distant metastases on CT scan of thorax and abdomen
* prior chemo- or antibody therapy
* history of significant cardiac disease
* current uncontrolled hypertension
* known hypersensitivity to the components of trastuzumab, pertuzumab, cisplatin, 5-follow-up or capecitabine
* known dihydropyrimidine dehydrogenase (DPD) deficiency
* ongoing or concomitant use of the antiviral drug sorivudine or its chemically related analogs, such as brivudine
* chronic treatment with high-dose intravenous corticosteroids
* previous malignancy within the last 5 years, with the exception of adequately treated cervical carcinoma in situ, localized non-melanoma skin cancer, or other curatively treated cancer without impact on the patient's overall prognosis according to the judgment of the investigator.
* psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Near Complete Pathological Response Rate | After 3 cycles (21 days) of neoadjuvant chemotherapy
  To increase the major pathological response rate (< 10% vital tumor cells) to neoadjuvant treatment by integrating both trastuzumab and pertuzumab into perioperative chemotherapy for HER-2 positive, resectable gastric cancer.

SECONDARY OUTCOMES:
Locoregional failure | At the time of surgery and at 5 years
R0 resection rate | At the time of surgery
Distant failure | At the time of surgery and at 5 years
Progression-free survival | 5 years after LPI
Recurrence-free survival | 5 years after LPI
Overall survival | 5 years after LPI
Toxicity | 5 years after LPI

CONTACTS AND LOCATIONS:
Overall Officials: Anna Dorothea Wagner, MD, Study Chair — Centre hospitalier universitaire vaudois, Lausanne
Locations (45):
- University Hospital Gent, Ghent, Flanders, Belgium
- North Estonia Medical Centre, Tallinn, Estonia
- France (5):
  - CHRU de Besancon - Hopital Jean Minjoz, Besançon
  - CHRU de Lille - Hopital Huriez, Lille
  - CHU de Bordeaux - Group Hospitalier Sud - Hopital Haut-Lévêque, Pessac
  - CHU de Reims - Hôpital Robert Debré, Reims
  - Institut Gustave Roussy, Villejuif
- Germany (11):
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Kliniken Essen-Mitte - Evang. Huyssens-Stiftung, Essen
  - Universitaetsmedizin Goettingen - Georg-August Universitaet, Göttingen
  - Asklepios Kliniken GmbH - Asklepios Klinik Barmbek, Hamburg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Onkologische Unter-Ems (Leer-Papenburg-Emden), Leer
  - Universitaetsklinikum Leipzig, Leipzig
  - Johannes Gutenberg Universitaetskliniken - Mainz University Medical Center, Mainz
  - Ludwig-Maximilians-Universitaet München - Campus Grosshadern, München
  - Technische Universität München - Klinikum Rechts der Isar, München
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Netherlands (2):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Academisch Medisch Centrum - UMC Universiteit van Amsterdam - site: VUMC, Amsterdam
- Oslo University Hospital - Radiumhospitalet, Oslo, Norway
- Portugal (2):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, Lisbon
  - Instituto Portugues De Oncologia - Centro Do Porto, Porto
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (6):
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hallym University Sacred Heart Hospital, Seoul
  - Severance Hospital YUCM, Seoul
  - Severance Hospital, Yonsei University Health System (YUCM), Seoul
  - The Catholic University of Korea-St. Vincent's Hospital, Suwon-Si Gyeonggi-do
- Spain (6):
  - Institut Catala d'Oncologia - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - ICO Badalona (Institut Catala d'Oncologia) - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebron - Institut Oncologia, Barcelona
  - ICO Girona - Hospital Dr Josep Trueta (Institut Catala d'Oncologia), Girona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico Universitario De Valencia, Valencia
- Switzerland (2):
  - Hôpitaux Universitaires de Genève - HUG, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- United Kingdom (4):
  - University Hospitals Birmingham NHS - UHB-Queen Elisabeth MC, Birmingham
  - University College London Hospitals (UCLH) - NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital - site: Sutton, Surrey, Sutton

REFERENCES:
- [Derived] Wagner AD, Grabsch HI, Mauer M, Marreaud S, Caballero C, Thuss-Patience P, Mueller L, Elme A, Moehler MH, Martens U, Kang YK, Rha SY, Cats A, Tokunaga M, Lordick F. EORTC-1203-GITCG - the "INNOVATION"-trial: Effect of chemotherapy alone versus chemotherapy plus trastuzumab, versus chemotherapy plus trastuzumab plus pertuzumab, in the perioperative treatment of HER2 positive, gastric and gastroesophageal junction adenocarcinoma on pathologic response rate: a randomized phase II-intergroup trial of the EORTC-Gastrointestinal Tract Cancer Group, Korean Cancer Study Group and Dutch Upper GI-Cancer group. BMC Cancer. 2019 May 24;19(1):494. doi: 10.1186/s12885-019-5675-4. PMID 31126258
- [Derived] Integration of Trastuzumab, with or without Pertuzumab, into Perioperative Chemotherapy of HER2- Positive Stomach Cancer: The INNOVATION Trial (EORTC-1203-GITCG). Oncol Res Treat. 2016;39(3):153-4; discussion 155. doi: 10.1159/000444702. No abstract available. PMID 27486629